CLINICAL TRIAL: NCT05952973
Title: The Impact of Online Educator Mircoskill Training and Parent Microskill Training on Student Sexual-Health Related Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashley Philliber (Other)
Responsible Party: Sponsor-Investigator, Ashley Philliber, Managing Director, Philliber Research & Evaluation
Organization: Philliber Research & Evaluation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Philliberdfusionparent
Record Dates: First submitted 2023-07-05; First posted 2023-07-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: HIV/AIDS Prevention; STI Prevention; Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SkillTalk (Experimental): Educators in the treatment group will receive access to an online educator microskill training platform. Parents/caregivers of students in the educators' classes will be assigned to treatment and receive access to a parent-specific online educator microskill training platform. Students in this group will receive "business as usual."
  Interventions: Behavioral: SkillTalk
- Business as usual (No Intervention): Business as usual.

INTERVENTIONS:
Behavioral: SkillTalk — Online Educator Mircoskill Training and Parent Microskill Training
  Other Names: SkillFlix
  Arms: SkillTalk

SUMMARY:
The goal of this clinical trial is to evaluate the impact of SkillTalk among educators, parents, and students. The main question[s] it aims to answer are:

* What is the impact of SkillTalk on student sexual-health related outcomes?
* What is the impact of SkillTalk on educator microskills?

Educator participants will use an online microskills training platform for one week. Parent participants will be asked to use a parent-specific online microskills training platform for one week. Youth participants will not be asked to do anything outside of "business as usual." Researchers will compare the treatment groups to the control groups to measure the impact of SkillTalk.

ELIGIBILITY:
Inclusion Criteria for Educators:

* Have fewer than three years teaching
* Teach youth in a class with at least 8 students
* Be able to obtain supervisor's or administration permission before beginning study
* Agree to be in compliance with district/school regulations about teaching sexual health and participating in a research study
* Agree to administer the assent/consent forms and student surveys.\

Inclusion Criteria for Students:

* Being in class of teacher who has agreed to participate
* Parental consent
* Assent to participate

Inclusion Criteria for Parents:

* Be the parent/guardian of a youth who has assented to participate
* Consent to their youth's participation
* Consent to view SkillTalk Parent site
* Need to speak English or Spanish
* Access to internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Condom knowledge | 1 month
  Students in the intervention group will show greater condom knowledge than students in the comparison group. This will consist of a scale that will be knowledge questions specific to the steps of condom usage. An overall score will be based on the percent correct. A higher score would be a more positive outcome.
Condom use | 1 month
  Students in the intervention group will show greater condom use self-efficacy than students in the comparison group. This will consist of a scale created for this study. This will be a self-efficacy scale using a 4-point strongly agree to strongly disagree scale. For each of these a higher score would be a more positive outcome.
STI knowledge | 1 month
  Students in the intervention group will show greater knowledge on STIs than students in the comparison group. This will be based on knowledge questions specific to the information found in SkillTalk. An overall score will be based on the percent correct. A higher score would be a more positive outcome.
Connectedness | 1 month
  Students in the intervention group will report greater feelings of connectedness with/perceived personalization of sexual health lesson messages than students in the comparison group. This will be based on a four point strongly agree to strongly disagree scale with questions specific to the information found in SkillTalk. An overall score will be based on the mean overall score of these questions. A higher score would be a more positive outcome.

SECONDARY OUTCOMES:
Self-efficacy and comfort with microskills | 1 month
  Educators in the intervention group will report greater self-efficacy and comfort with condom and STI Microskills than educators in the comparison group. This will be based on a four point strongly agree to strongly disagree scale with questions specific to the information found in SkillTalk. An overall score will be based on the mean overall score of these questions. A higher score would be a more positive outcome.
Student impressions of educator skills | 1 month
  Students in the intervention group will report more positive perceptions of educator knowledge, skill, and comfort to teach sexual health lessons. This will be based on a four point strongly agree to strongly disagree scale with questions specific to the information found in SkillTalk. An overall score will be based on the mean overall score of these questions. A higher score would be a more positive outcome.
Frequency of parent-child communication | 1 month
  Parents in the intervention group will report more frequent communication about sexual health with their youth. This will be based on a scale that will include daily, more than twice a week, twice per week, weekly, bi weekly, monthly, less than monthly, and never. A greater frequency of communication would be a more positive outcome.
Comfort in parent-child communication | 1 month
  Parents in the intervention group will report more comfort in communicating with their child about sexual health. This will be based on a four point strongly agree to strongly disagree scale with questions specific to the information found in SkillTalk. An overall score will be based on the mean overall score of these questions. A higher score would be a more positive outcome.
Parent-child communication | 1 month
  Parents in the intervention group will be perceived as better communicators by their children. This will be based on a four point strongly agree to strongly disagree scale with questions specific to the information found in SkillTalk. An overall score will be based on the mean overall score of these questions. A higher score would be a more positive outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Philliber Research & Evaluation, Accord, New York, United States

IPD SHARING:
Plan to Share IPD: No